CLINICAL TRIAL: NCT03201692
Title: Improving Dynamic Balance and Gait Adaptability Using Treadmill Training With Visual Cues in Subjects With Neurological Disorders: Design of a Pilot Study
Brief Title: Improving Dynamic Balance and Gait Adaptability Using Treadmill Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Davide Cattaneo, Research Coordinator, LaRiCE Lab, PhD, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT02960984UL_SM
Record Dates: First submitted 2017-06-09; First posted 2017-06-28 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis; Stroke; Parkinson Disease
MeSH Terms: conditions — Multiple Sclerosis; Stroke; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treadmill Training (Active Comparator): 40' treadmill training walking holding the handrail
  Interventions: Device: Treadmill training
- Virtual Reality Treadmill Training (Experimental): 40' treadmill training walking with virtual visual and auditory cues
  Interventions: Device: Virtual Reality Treadmill Training

INTERVENTIONS:
Device: Virtual Reality Treadmill Training — Subjects in the experimental group will receive 40 minutes comprising exercises focused on improving dynamic balance following auditory and visual cues.
  Other Names: C-mill treadmill
  Arms: Virtual Reality Treadmill Training
Device: Treadmill training — Subjects in the active comparator group will receive 40 minutes walking training aimed to improve velocity and endurance.
  Arms: Treadmill Training

SUMMARY:
Balance and gait problems in subjects with neurological disease lead to reduced mobility, loss of independence and frequent falls. Treadmill training is a widely used form of treatment and it has been used in subjects with neurological disease to ameliorate walking and balance deficits. The Virtual Reality Treadmill as a therapeutic tool has been recently introduced to practice gait adaptability elicited by aligning foot placement relative to the projected visual context.

Forty-eight subjects with neurological disease will receive treadmill training treatment randomly divided in Traditional Treadmill training and Virtual Reality Treadmill training.

The aim of this randomized controlled study is to assess whether Treadmill training with Virtual Reality is better than Traditional Treadmill training in improving dynamic balance and cognitive aspects in subjects with neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis (no relapse within the previous three months;), Parkinsons Disease (Hoenhn and Yahr Scale ≤4), Stroke (Time from onset >2 months)
* Able to walk 20 meters with or without assistive device
* Cognitive impairment (MMSE score ≥ 21)

Exclusion Criteria:

* Unable to understand the aim of the study and unable to sign the informed consent
* Steroidal drugs therapy for subjects with Multiple Sclerosis
* Subjects with Psychiatric disorders
* Subjects with Visual impairments
* Subjects with cardiovascular disease

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-04-10 (Estimated); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in the Modified Dynamic Gait Index | Change from Baseline Modified Dynamic Gait Index scores at 3-5 weeks
  Tool used to assess dynamic balance
Change in the 6 minutes walking test | Change from Baseline 6 minutes walking test scores at 3-5 weeks
  tool used to assess walking endurance

SECONDARY OUTCOMES:
Change in Activity Balance Confidence | Change from Baseline Activity Balance Confidence scores at 3-5 weeks
  Tool used to assess of balance confidence in daily life activities
Change in 10-meter walking test | Change from Baseline10-meter walking test scores at 3-5 weeks
  Tool used to assess walking speed in 3 different conditions ( normal speed, fastest speed, cognitive dual task)
Change in Trial Making test | Change from Baseline Trial Making test scores at 3-5 weeks
  The Trail Making Test is a neuropsychological tapping visual attention and task switching. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
Change in Raven's Matrices | Change from Baseline Raven's Matrices scores at 3-5 weeks
  Test used in measuring abstract reasoning and regarded as a non-verbal estimate of fluid intelligence.

CONTACTS AND LOCATIONS:
Locations (1):
- Don Gnocchi Foundation, Milan, Italy

IPD SHARING:
Plan to Share IPD: No